CLINICAL TRIAL: NCT04503083
Title: A Multidisciplinary Approach to the Identification of BIOmarkers of MIGraine: a Proof of Concept Study Based on the Stratification of Responders to CGRP Monoclonal Antibodies
Brief Title: BIOmarkers of MIGraine: a Proof of Concept Study Based on the Stratification of Responders to CGRP Monoclonal Antibodies
Acronym: BIOMIGA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Other Study IDs: BIOMIGA2020
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2020-07

CONDITIONS: Migraine
Keywords: Migraine; Biomarkers; CGRP monoclonal Antibodies
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for DNA extraction for DNA methylation analysis and for CGRP-related polymorphisms, and for biochemical profiling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Migraine patients: * Excellent responder, a patient who experiences a >75% decrease of either the monthly number of migraine days or the monthly number of moderate/severe headache days during the last 4 weeks of treatment as compared to baseline;
  * Responder, a patient who experiences a >50% decrease of either the monthly number of migraine days or the monthly number of moderate/severe headache days during the last 4 weeks of treatment as compared to baseline;
  * Non responder, a patient who experiences a decrease of either the monthly number of migraine days or the monthly number of moderate/severe headache days ranging from 26 to 49% during the last 4 weeks of treatment as compared to baseline;
  * Full non responder, a patient who experiences a <25% decrease of either the monthly number of migraine days or the monthly number of moderate/severe headache days during the last 4 weeks of treatment as compared to baseline.

SUMMARY:
Migraine is the 2nd most disabling neurological disease. It affects 14.7% of the population (children and adults) of whom 80% are female. In the European Union, the total annual cost of migraine is of 111 billion euros. If not adequately treated, migraine can evolve into the more severe chronic form (CM), defined by >15 headache days/month, where burden and costs increase exponentially.

Until very recently, available preventive treatments for migraine were non-specific, of limited efficacy and scarce tolerability. In 2018, monoclonal antibodies (mABs) against calcitonin gene-related peptide (CGRP) receptor have been approved. Since CGRP is one of the main modulators of the trigeminal system, mABs against CGRP are the first specific preventive treatment for migraine ever developed. They are highly effective in a subgroup of patients, well tolerated, but costly.

In this frame, the main objective of BIOMIGA project is to identify predictive biomarkers of response to CGRP-mABs in patients with severe forms of migraine. To this end, the investigators will use an integrated hypothesis-based and data-driven, multidisciplinary approach that combines' omic testing in a deep-phenotyped migraine population and parallel fundamental research in a validated animal model of migraine. Three partners, Headache Science Centre, IRCCS C. Mondino Foundation, University of Pavia, Italy, Headache Research Group Vall d'Hebron Institute of Research, Barcelona, Spain and Institut für Systemische Neurowissenschaften, Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany with an established long-standing and complementary expertise in neuroimaging, biochemical profiling and epigenetics in humans and in animal modeling of migraine will collaborate to achieve the Project's objective.

The investigators expect important spin-offs to the improved management of migraine, both in terms of increased efficacy and cost saving, but also to understand CGRP-based mechanisms underlying migraine pathophysiology and to set the basis for a pathophysiologically driven classification. Healthcare providers and the pharmaceutical industry will be engaged once the biomarker(s) have been identified to optimize access to care and the use of resource, as well as to reduce disability and socio-economic impact of migraine.

DETAILED DESCRIPTION:
Almost 15% of European citizens suffer from migraine and its comorbidities. Migraine is the second most disabling chronic neurological disease, with devastating repercussions on the life of those who are affected, their relatives and society. Migraine manifests in recurring attacks lasting 4-72 hours characterized by severe head pain, often throbbing, associated with nausea, photo and phonophobia, vomiting, cognitive deficits, severe emotional distress and complete disability. If not diagnosed and appropriately treated, migraine can transform into a chronic form (15 or more days of headache/ month) often associated with acute medication overuse and severe comorbidities such as depression, anxiety and panic disorders.

The disability associated to migraine is closely related to the frequency of the attacks. Epidemiological studies show that in Europe 34$ of migraineurs suffer from more than 5 headache days per month and 1-3% of the general population has migraine on more than 15 days/month, thus qualifying for the diagnosis of Chronic Migraine (CM).

Migraine is a genetically-driven, chronic "neurosensorial" disorder, where the unpredictable recurrence of the attacks is modulated by the variable efficiency of the fine-tuned interplay of the brain with dynamic sensory stimuli originating from the internal or external environment.

Migraine can be viewed as a cycling functional disorder that affects several areas of the brain, involving multiple pathways ultimately leading to the excessive activation of trigeminovascular afferents in the meninges with the local release of vasoactive substances (calcitonin gene-related peptide - CGRP ) and the activation of the neuroinflammatory cascade.

Unlike several other chronic neurological diseases, migraine can be successfully treated and prevented. Unfortunately, this is true only for subgroups of patients and for a limited period, due to the nonspecific therapeutic armamentarium available: calcium antagonists, beta-blockers, antidepressants, antiepileptics and, only for chronic migraine, onabotulinumtoxin-A. This is the direct consequence of the complex pathophysiology of the disease, but mostly and, more importantly, by the total absence of biomarkers of disease and of responsiveness to available drugs.

In the last years, enormous efforts have indeed been undertaken to identify biomarker of migraine, especially for the chronic form. Functional imaging has provided important clues on the machinery underlying attack generation and imaging biomarkers for chronic migraine, whereas it has become evident that epigenetic processes - DNA methylation in particular - may play an important role in the phenotypical expression of migraine. Attack recurrence and the associated changes in neuronal activity may indeed cause epigenetic changes that alter synaptic plasticity, thus leading to more frequent migraine attacks and ultimately promotes stable epigenetic changes in a feed-forward loop. Circulating levels of CGRP have also been evaluated as a possible peripheral biomarker of migraine in consideration of the seminal observations that CGRP levels increase in the external jugular vein during a migraine attack.

The second half of 2018 marked a revolution in the treatment of migraine: the advent of the monoclonal antibodies (mABs) directed against CGRP or its receptor. They proved safe and effective in reducing migraine frequency and represent the first class of preventive drugs targeting a specific step in the cascade of events leading to the migraine attack. Results from clinical trials have shown that approximately 1/3 of patients are excellent responders (>75% reduction in headache days) whilst 1/3 patients are non- or poor responders (<25% reduction in headache days) to CGRP-targeted mABs.

CGRP-targeted mABs do not interfere with other systems or medications. Consequently, the fact that patients can be stratified as responders and non-responders creates a unique opportunity to better understand the difference of response in patients clinically alike and, through this, provide unprecedented insights into the pathophysiology of migraine allowing the migraine field to move towards a pathophysiological driven classification.

For decades the migraine scientific community has been searching for biomarkers associated with the disease or with its response to treatment. Unfortunately, to date none has been validated. This failure is likely related to multiple reasons: the complex and dynamic nature of migraine-associated biological processes (attack vs. pre-post interictal phase), the multiplicity of neurotransmitters (serotonin dopamine, neuropeptides, etc.), the neuroanatomical structures (peripheral, central) and the interindividual variability of disease expression. Moreover, the reasons for the failure of previous studies are also associated with the variability between studies, in terms of methodology, population and endpoints, which has led to inconsistent findings and low estimate precision.

Now, a selective class of preventive drugs that specifically target a biological step in migraine disease has become available, prompting the possibility to precisely stratify migraine subjects on the basis of their pharmacological response. The availability of high-throughput technologies is providing unprecedented opportunities to identify molecular markers of complex disease by extracting meaningful signatures from complex and heterogeneous sets of data. Molecular biomarkers of thoroughly stratified populations can be combined with deep clinical phenotyping and also with epigenetic, pharmacogenetic and neuroimaging variables, that are relevant for migraine. The availability of migraine-specific animal models also contributes to identifying and firmly placing important pieces to the migraine puzzle.

Against this background, a hybrid data-driven and knowledge-based approach building on clinical and preclinical inputs and including phenotype, genetic, neuroimaging and animal data will provide a large informative dataset that can be effectively analyzed with machine and deep learning algorithms for feature selection, modeling and for subsequent cross-validation to ultimately yield a precise, robust and reproducible model for predicting the response of migraine to a specifically targeted preventive treatment. This will be a crucial step in the therapeutic decision process, especially in the most severe and disabling form of migraine, chronic migraine. It will also provide additional positive implications in the field, such as prompting the ground for a pathophysiology-driven diagnosis and, equally important, robust scientific evidence to European decision makers and health-care providers for optimizing the distribution of resources and rationalizing the access to care of migraine sufferers. Engagement of patients is envisaged both in the planning and conducting of the study to ensure that project methodology and results are in line with their needs and expectations, thus favoring the translation into clinical practice.

Monoclonal antibodies targeting CGRP (CGRP-mABs) have been shown to be effective in the preventive treatment of migraine. They are large molecules that do not cross the blood brain barrier, have a long half-life (20-45 days) and do not interact pharmacologically. They are administered parenterally, which warrants less intra-individual variations and a better adherence to treatment.

CGRP-mABs have proven safe and effective in multiple phase II and III randomized controlled clinical trials and were approved by FDA and European Medicines Agency (EMA) as a preventive treatment for migraine. Four CGRP-mABs have been studied and 3 of them have been approved by EMA in late 2018 and 2019: erenumab, galcanezumab and fremanezumab.

A strong body of evidence suggests that CGRP-mABs induce a 50% response (50% reduction in monthly headache days) in about 50% of subjects, with a 75% response in 30-40% of patients. The latter group, from now on defined as 'excellent responders', represents an interesting subgroup of migraine subjects whose disease is likely particularly dependent on CGRP-related pathways. Hence, the availability of mABs targeting CGRP together with the demonstration of their efficacy in relevant subgroups of subjects prompt a formidable tool to tackle precisely a subset of mechanisms and pathways underlying the disease.

CGRP-targeted mABs do not interfere with other systems or medications. Consequently, the fact that patients can be precisely stratified as excellent responders and non-responders creates a unique novel opportunity to unravel hitherto concealed differences between patients with the same diagnosis and, through this, provides unprecedented insights into the pathophysiology of migraine. Ultimately, this will allow the migraine field to move towards a neurobiological definition of responders and a pathophysiological driven classification. Defining predictors to this response will in turn allow obtaining a more cost-effective approach to migraine healthcare. Engagement of patients is envisaged both in the planning and conducting of the study based on the long-standing collaboration with the European Migraine and Headache Alliance (EMHA), which has been aligned and involved in the preparation of the present proposal.

Epigenetics is acquiring an increasing importance in the panorama of biological events that leads to the transformation of episodic migraine (EM) into chronic migraine (CM). Frequent recurrence of migraine attacks may indeed promote stable epigenetic changes in a feed-forward loop thus altering synaptic plasticity. So far, the most significant associated CpG sites related to migraine chronification are SH2D5, NPTX2 and RAMP1, three brain-expressed genes involved in the regulation of synaptic plasticity and CGRP modulation. However, it is still not known whether a specific profile of DNA methylation, which is a stable epigenetic chemical marker crucial for many cellular activities, can predict the clinical response to preventive therapy in migraine patients.

Neuroimaging Functional imaging studies have revolutionized this area and provided unique neuroanatomical and functional insights into migraine machinery. Functional imaging has revealed that the pathophysiology of migraine crucially involves hypothalamo-thalamo-brainstem networks. Pharmacological imaging has begun to shed light on how medications may enfold their effect in migraine.

The combination of structural and functional imaging parameters with and without external input will give us the unique opportunity to characterize patients who respond to CGRP_targeting antibodies against those who do not. These data will then be an additional powerful source for informing animal projects and also machine learning algorithms.

The overarching and main objective of this proposal is the identification of predictive biomarkers of response to treatment with CGRP-targeted mAbs in chronic migraine, the most severe and disabling form of migraine.

Screening will be performed at visit 1 (month 0). Patients will sign the informed consent and will be instructed to fill in a headache diary and will return after 1 month (+2 days) for visit 2 (V2). At V2, after verification of inclusion/exclusion criteria, enrolled subjects will fill in the protocol scales (Assessment of disability - monthly MIDAS, Headache Impact Test 6 (HIT-6) -, depression - Beck Depression Inventory, BDI-II -, anxiety - Beck Anxiety Inventory, Beck Anxiety Inventory (BAI) -, quality of life - MSQ- , subjective cognitive impairment scale for migraine attacks - Mig-SCog -, comorbidities, acute medications intake, anxiety and depression - Beck scales - and Emergency Room Use), they will undergo blood sampling, neuroimaging and they will receive the first treatment administration.

Healthy controls will be screened at V1 and, following the verification of the satisfaction of inclusion/exclusion criteria and the signature of the informed consent, will fill in the protocol scale, they will undergo blood sampling and neuroimaging.

The first dose (defined according to the indication approved by the Local Health Authorities) of the CGRP-targeting monoclonal antibody will be administered during the hospital visit.

The patient will receive 2 additional doses of the drug and a training on the modality of self-injection and specific indication of the day they will perform the self-injection. They will also receive the headache diary and associated instructions for filling it in regularly during the following 3 months.

No drug treatment is foreseen for healthy controls.

No concomitant migraine preventive treatment will be allowed during the screening, baseline and the 3-month treatment period.

Abortive medications will be allowed, but the type and formulation should be kept stable during the study. Data about their doses and frequencies will be recorded.

A remote visit will be scheduled 30 (week 4) and 60 (week 8) days after day 1 to monitor patient's health status, remind the treatment schedule and collect the data from the headache diaries (visit 3 and 4).

At visit 5 (week 12), all migraine subjects will undergo:

* Assessment of disability (MIDAS, HIT-6), work impairment (WPAI scale), evaluation of acute medications intake, anxiety and depression, quality of life (MSQ), Emergency Room Use.
* Assessment of treatment efficacy through the headache diaries (migraine days/month)
* Assessment of treatment satisfaction with validated patient reported outcomes (PROs).

Excellent responders and non-responders will also undergo neuroimaging evaluation: 3Tesla Magnetic resonance imaging (MRI) involving Structural (sMRI) resting state MRI (rsMRI), Arterial Spin Labelling (ASL) and Diffusion Tensor Imaging (DTI).

ELIGIBILITY:
Inclusion Criteria:

Migraine patients

* Adults between 25 and 55 years of age of both gender;
* European background;
* Patients diagnosed with high-frequency migraine (HFM) 8 or more migraine days days/month) or CM with or without aura (>15 headache days migraine/month, of which 8 have migraine characteristics) according to the International Classification of Headache Disorders, 3rd edition, (ICHD-3);
* Females have to be postmenopausal for at least one year, surgically sterile or otherwise incapable of pregnancy, or using an acceptable method of birth control.

Healthy controls

* Adults between 25 and 55 years of age of both genders;
* European background;
* Absence of any past or first-degree familial history of recurrent primary or secondary headache disorders.

Exclusion Criteria:

For the clinical population:

* Headache on more than 25 days/month in the last 3 months;
* Medication overuse according to the ICHD-3 criteria.

For the entire study population (migraine and healthy controls)

* Presence of any other significant medical condition (neurological disorders, severe psychiatric illness or cardiovascular disease);
* Evidence of drug, smoking or alcohol abuse or dependence within 12 months prior to V1, based on medical records or patient self-report. An alcohol consumption >100mg/week will be considered an abuse;
* Pregnant or breastfeeding women;
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant who are not on contraception;
* Concomitant use of other migraine preventive drugs that may interfere with the endpoints of the study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Migraine patients and Healthy controls.
  The Health controls will be recruited among hospital staff and non-related acquaintances of the patients.
  All patients enrolled in the study will be treated with CGRP-targeting mABs according to the indications approved by their National regulatory bodies
Sampling Method: Non-Probability Sample
Enrollment: 219 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Biomarkers and CGRP-targeting mABs | Day 0 and Week 12
  To identify a computational algorithm using a machine learning approach based on different types of biomarkers (demographic, clinical, psychological, cognitive, epigenetic, pharmacogenetic, biochemical and structural & functional brain imaging) that is predictive of response to the class of the CGRP-targeting mABs.

SECONDARY OUTCOMES:
Methylation levels | Day 0 and Week 12
  Difference in methylation levels in migraine subjects as compared to healthy controls
Brain morphometric measures | Day 0 and Week 12
  Differences in brain morphometric measures between migraine patients and healthy controls at the neuroanatomic and neurofunctional levels
Pharmacogenetic, biochemical, clinical and psychological markers | Day 0 and Week 12
  Differences in pharmacogenetic, biochemical, clinical and psychological markers between migraine patients and healthy controls
Methylation levels at the neuroanatomic and neurofunctional levels | Day 0 and Week 12
  Difference in methylation levels in migraine subjects between migraine patients and healthy controls at the neuroanatomic and neurofunctional levels
Morphometric measures | Day 0 and Week 12
  Differences in brain morphometric measures between migraine subjects who are responder and those who are non responders to CGRP-targeting mABs
Pharmacogenetic, biochemical, clinical and psychological markers in responder and non responders | Day 0 and Week 12
  Differences in pharmacogenetic, biochemical, clinical and psychological between migraine subjects who are responder and those who are non responders to CGRP-targeting mABs

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Tassorelli, Prof, Principal Investigator — IRCCS Mondino Foundation, Pavia
Locations (3):
- Institut für Systemische Neurowissenschaften, Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany
- Headache Science Center, Pavia, Italy
- Headache Research Group Vall d'Hebron Institute of Research, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steiner TJ, Stovner LJ, Vos T. GBD 2015: migraine is the third cause of disability in under 50s. J Headache Pain. 2016 Dec;17(1):104. doi: 10.1186/s10194-016-0699-5. Epub 2016 Nov 14. No abstract available. PMID 27844455
- [Background] Steiner TJ, Jensen R, Katsarava Z, Linde M, MacGregor EA, Osipova V, Paemeleire K, Olesen J, Peters M, Martelletti P. Aids to management of headache disorders in primary care (2nd edition) : on behalf of the European Headache Federation and Lifting The Burden: the Global Campaign against Headache. J Headache Pain. 2019 May 21;20(1):57. doi: 10.1186/s10194-018-0899-2. PMID 31113373
- [Background] May A, Schulte LH. Chronic migraine: risk factors, mechanisms and treatment. Nat Rev Neurol. 2016 Aug;12(8):455-64. doi: 10.1038/nrneurol.2016.93. Epub 2016 Jul 8. PMID 27389092
- [Background] Goadsby PJ, Holland PR, Martins-Oliveira M, Hoffmann J, Schankin C, Akerman S. Pathophysiology of Migraine: A Disorder of Sensory Processing. Physiol Rev. 2017 Apr;97(2):553-622. doi: 10.1152/physrev.00034.2015. PMID 28179394
- [Background] Conti P, D'Ovidio C, Conti C, Gallenga CE, Lauritano D, Caraffa A, Kritas SK, Ronconi G. Progression in migraine: Role of mast cells and pro-inflammatory and anti-inflammatory cytokines. Eur J Pharmacol. 2019 Feb 5;844:87-94. doi: 10.1016/j.ejphar.2018.12.004. Epub 2018 Dec 6. PMID 30529470
- [Background] Schulte LH, May A. Functional Neuroimaging in Migraine: Chances and Challenges. Headache. 2016 Oct;56(9):1474-1481. doi: 10.1111/head.12944. Epub 2016 Sep 22. PMID 27654831
- [Background] Schulte LH, Allers A, May A. Hypothalamus as a mediator of chronic migraine: Evidence from high-resolution fMRI. Neurology. 2017 May 23;88(21):2011-2016. doi: 10.1212/WNL.0000000000003963. Epub 2017 Apr 26. PMID 28446645
- [Background] Gerring ZF, McRae AF, Montgomery GW, Nyholt DR. Genome-wide DNA methylation profiling in whole blood reveals epigenetic signatures associated with migraine. BMC Genomics. 2018 Jan 22;19(1):69. doi: 10.1186/s12864-018-4450-2. PMID 29357833
- [Background] Zagami AS, Goadsby PJ, Edvinsson L. Stimulation of the superior sagittal sinus in the cat causes release of vasoactive peptides. Neuropeptides. 1990 Jun;16(2):69-75. doi: 10.1016/0143-4179(90)90114-e. PMID 2250767
- [Background] Edvinsson L, Haanes KA, Warfvinge K, Krause DN. CGRP as the target of new migraine therapies - successful translation from bench to clinic. Nat Rev Neurol. 2018 Jun;14(6):338-350. doi: 10.1038/s41582-018-0003-1. PMID 29691490
- [Background] Raffaelli B, Reuter U. The Biology of Monoclonal Antibodies: Focus on Calcitonin Gene-Related Peptide for Prophylactic Migraine Therapy. Neurotherapeutics. 2018 Apr;15(2):324-335. doi: 10.1007/s13311-018-0622-7. PMID 29616494
- [Background] Ferroni P, Barbanti P, Della-Morte D, Palmirotta R, Jirillo E, Guadagni F. Redox Mechanisms in Migraine: Novel Therapeutics and Dietary Interventions. Antioxid Redox Signal. 2018 Apr 20;28(12):1144-1183. doi: 10.1089/ars.2017.7260. Epub 2017 Nov 21. PMID 28990418
- [Background] Demartini C, Greco R, Zanaboni AM, Sances G, De Icco R, Borsook D, Tassorelli C. Nitroglycerin as a comparative experimental model of migraine pain: From animal to human and back. Prog Neurobiol. 2019 Jun;177:15-32. doi: 10.1016/j.pneurobio.2019.02.002. Epub 2019 Feb 13. PMID 30771365
- [Background] Kambur O, Kaunisto MA, Winsvold BS, Wilsgaard T, Stubhaug A, Zwart JA, Kalso E, Nielsen CS. Genetic variation in P2RX7 and pain tolerance. Pain. 2018 Jun;159(6):1064-1073. doi: 10.1097/j.pain.0000000000001188. PMID 29470314
- [Background] Brainstorm Consortium; Anttila V, Bulik-Sullivan B, Finucane HK, Walters RK, Bras J, Duncan L, Escott-Price V, Falcone GJ, Gormley P, Malik R, Patsopoulos NA, Ripke S, Wei Z, Yu D, Lee PH, Turley P, Grenier-Boley B, Chouraki V, Kamatani Y, Berr C, Letenneur L, Hannequin D, Amouyel P, Boland A, Deleuze JF, Duron E, Vardarajan BN, Reitz C, Goate AM, Huentelman MJ, Kamboh MI, Larson EB, Rogaeva E, St George-Hyslop P, Hakonarson H, Kukull WA, Farrer LA, Barnes LL, Beach TG, Demirci FY, Head E, Hulette CM, Jicha GA, Kauwe JSK, Kaye JA, Leverenz JB, Levey AI, Lieberman AP, Pankratz VS, Poon WW, Quinn JF, Saykin AJ, Schneider LS, Smith AG, Sonnen JA, Stern RA, Van Deerlin VM, Van Eldik LJ, Harold D, Russo G, Rubinsztein DC, Bayer A, Tsolaki M, Proitsi P, Fox NC, Hampel H, Owen MJ, Mead S, Passmore P, Morgan K, Nothen MM, Rossor M, Lupton MK, Hoffmann P, Kornhuber J, Lawlor B, McQuillin A, Al-Chalabi A, Bis JC, Ruiz A, Boada M, Seshadri S, Beiser A, Rice K, van der Lee SJ, De Jager PL, Geschwind DH, Riemenschneider M, Riedel-Heller S, Rotter JI, Ransmayr G, Hyman BT, Cruchaga C, Alegret M, Winsvold B, Palta P, Farh KH, Cuenca-Leon E, Furlotte N, Kurth T, Ligthart L, Terwindt GM, Freilinger T, Ran C, Gordon SD, Borck G, Adams HHH, Lehtimaki T, Wedenoja J, Buring JE, Schurks M, Hrafnsdottir M, Hottenga JJ, Penninx B, Artto V, Kaunisto M, Vepsalainen S, Martin NG, Montgomery GW, Kurki MI, Hamalainen E, Huang H, Huang J, Sandor C, Webber C, Muller-Myhsok B, Schreiber S, Salomaa V, Loehrer E, Gobel H, Macaya A, Pozo-Rosich P, Hansen T, Werge T, Kaprio J, Metspalu A, Kubisch C, Ferrari MD, Belin AC, van den Maagdenberg AMJM, Zwart JA, Boomsma D, Eriksson N, Olesen J, Chasman DI, Nyholt DR, Avbersek A, Baum L, Berkovic S, Bradfield J, Buono RJ, Catarino CB, Cossette P, De Jonghe P, Depondt C, Dlugos D, Ferraro TN, French J, Hjalgrim H, Jamnadas-Khoda J, Kalviainen R, Kunz WS, Lerche H, Leu C, Lindhout D, Lo W, Lowenstein D, McCormack M, Moller RS, Molloy A, Ng PW, Oliver K, Privitera M, Radtke R, Ruppert AK, Sander T, Schachter S, Schankin C, Scheffer I, Schoch S, Sisodiya SM, Smith P, Sperling M, Striano P, Surges R, Thomas GN, Visscher F, Whelan CD, Zara F, Heinzen EL, Marson A, Becker F, Stroink H, Zimprich F, Gasser T, Gibbs R, Heutink P, Martinez M, Morris HR, Sharma M, Ryten M, Mok KY, Pulit S, Bevan S, Holliday E, Attia J, Battey T, Boncoraglio G, Thijs V, Chen WM, Mitchell B, Rothwell P, Sharma P, Sudlow C, Vicente A, Markus H, Kourkoulis C, Pera J, Raffeld M, Silliman S, Boraska Perica V, Thornton LM, Huckins LM, William Rayner N, Lewis CM, Gratacos M, Rybakowski F, Keski-Rahkonen A, Raevuori A, Hudson JI, Reichborn-Kjennerud T, Monteleone P, Karwautz A, Mannik K, Baker JH, O'Toole JK, Trace SE, Davis OSP, Helder SG, Ehrlich S, Herpertz-Dahlmann B, Danner UN, van Elburg AA, Clementi M, Forzan M, Docampo E, Lissowska J, Hauser J, Tortorella A, Maj M, Gonidakis F, Tziouvas K, Papezova H, Yilmaz Z, Wagner G, Cohen-Woods S, Herms S, Julia A, Rabionet R, Dick DM, Ripatti S, Andreassen OA, Espeseth T, Lundervold AJ, Steen VM, Pinto D, Scherer SW, Aschauer H, Schosser A, Alfredsson L, Padyukov L, Halmi KA, Mitchell J, Strober M, Bergen AW, Kaye W, Szatkiewicz JP, Cormand B, Ramos-Quiroga JA, Sanchez-Mora C, Ribases M, Casas M, Hervas A, Arranz MJ, Haavik J, Zayats T, Johansson S, Williams N, Dempfle A, Rothenberger A, Kuntsi J, Oades RD, Banaschewski T, Franke B, Buitelaar JK, Arias Vasquez A, Doyle AE, Reif A, Lesch KP, Freitag C, Rivero O, Palmason H, Romanos M, Langley K, Rietschel M, Witt SH, Dalsgaard S, Borglum AD, Waldman I, Wilmot B, Molly N, Bau CHD, Crosbie J, Schachar R, Loo SK, McGough JJ, Grevet EH, Medland SE, Robinson E, Weiss LA, Bacchelli E, Bailey A, Bal V, Battaglia A, Betancur C, Bolton P, Cantor R, Celestino-Soper P, Dawson G, De Rubeis S, Duque F, Green A, Klauck SM, Leboyer M, Levitt P, Maestrini E, Mane S, De-Luca DM, Parr J, Regan R, Reichenberg A, Sandin S, Vorstman J, Wassink T, Wijsman E, Cook E, Santangelo S, Delorme R, Roge B, Magalhaes T, Arking D, Schulze TG, Thompson RC, Strohmaier J, Matthews K, Melle I, Morris D, Blackwood D, McIntosh A, Bergen SE, Schalling M, Jamain S, Maaser A, Fischer SB, Reinbold CS, Fullerton JM, Guzman-Parra J, Mayoral F, Schofield PR, Cichon S, Muhleisen TW, Degenhardt F, Schumacher J, Bauer M, Mitchell PB, Gershon ES, Rice J, Potash JB, Zandi PP, Craddock N, Ferrier IN, Alda M, Rouleau GA, Turecki G, Ophoff R, Pato C, Anjorin A, Stahl E, Leber M, Czerski PM, Cruceanu C, Jones IR, Posthuma D, Andlauer TFM, Forstner AJ, Streit F, Baune BT, Air T, Sinnamon G, Wray NR, MacIntyre DJ, Porteous D, Homuth G, Rivera M, Grove J, Middeldorp CM, Hickie I, Pergadia M, Mehta D, Smit JH, Jansen R, de Geus E, Dunn E, Li QS, Nauck M, Schoevers RA, Beekman AT, Knowles JA, Viktorin A, Arnold P, Barr CL, Bedoya-Berrio G, Bienvenu OJ, Brentani H, Burton C, Camarena B, Cappi C, Cath D, Cavallini M, Cusi D, Darrow S, Denys D, Derks EM, Dietrich A, Fernandez T, Figee M, Freimer N, Gerber G, Grados M, Greenberg E, Hanna GL, Hartmann A, Hirschtritt ME, Hoekstra PJ, Huang A, Huyser C, Illmann C, Jenike M, Kuperman S, Leventhal B, Lochner C, Lyon GJ, Macciardi F, Madruga-Garrido M, Malaty IA, Maras A, McGrath L, Miguel EC, Mir P, Nestadt G, Nicolini H, Okun MS, Pakstis A, Paschou P, Piacentini J, Pittenger C, Plessen K, Ramensky V, Ramos EM, Reus V, Richter MA, Riddle MA, Robertson MM, Roessner V, Rosario M, Samuels JF, Sandor P, Stein DJ, Tsetsos F, Van Nieuwerburgh F, Weatherall S, Wendland JR, Wolanczyk T, Worbe Y, Zai G, Goes FS, McLaughlin N, Nestadt PS, Grabe HJ, Depienne C, Konkashbaev A, Lanzagorta N, Valencia-Duarte A, Bramon E, Buccola N, Cahn W, Cairns M, Chong SA, Cohen D, Crespo-Facorro B, Crowley J, Davidson M, DeLisi L, Dinan T, Donohoe G, Drapeau E, Duan J, Haan L, Hougaard D, Karachanak-Yankova S, Khrunin A, Klovins J, Kucinskas V, Lee Chee Keong J, Limborska S, Loughland C, Lonnqvist J, Maher B, Mattheisen M, McDonald C, Murphy KC, Nenadic I, van Os J, Pantelis C, Pato M, Petryshen T, Quested D, Roussos P, Sanders AR, Schall U, Schwab SG, Sim K, So HC, Stogmann E, Subramaniam M, Toncheva D, Waddington J, Walters J, Weiser M, Cheng W, Cloninger R, Curtis D, Gejman PV, Henskens F, Mattingsdal M, Oh SY, Scott R, Webb B, Breen G, Churchhouse C, Bulik CM, Daly M, Dichgans M, Faraone SV, Guerreiro R, Holmans P, Kendler KS, Koeleman B, Mathews CA, Price A, Scharf J, Sklar P, Williams J, Wood NW, Cotsapas C, Palotie A, Smoller JW, Sullivan P, Rosand J, Corvin A, Neale BM, Schott JM, Anney R, Elia J, Grigoroiu-Serbanescu M, Edenberg HJ, Murray R. Analysis of shared heritability in common disorders of the brain. Science. 2018 Jun 22;360(6395):eaap8757. doi: 10.1126/science.aap8757. PMID 29930110
- [Background] Kroger IL, May A. Pharmacological neuroimaging in headache and pain. Curr Opin Neurol. 2013 Jun;26(3):254-61. doi: 10.1097/WCO.0b013e32836085df. PMID 23511443
- [Background] Wan D, Hou L, Zhang X, Han X, Chen M, Tang W, Liu R, Dong Z, Yu S. DNA methylation of RAMP1 gene in migraine: an exploratory analysis. J Headache Pain. 2015;16:90. doi: 10.1186/s10194-015-0576-7. Epub 2015 Oct 26. PMID 26501962